CLINICAL TRIAL: NCT04153318
Title: Comparing of FFOCT Imaging for Pancreatic Tissue Sample Obtained by EUSFNB and Conventional Histological Examination
Brief Title: Diagnostic Efficacy of FFOCT Imaging for Tissue Sample Obtained by EUSFNB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, chief of the Gastroenterology, Changhai Hospital
Other Study IDs: FFOCT
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Diseases
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: full-field optical coherence tomography — Pancreatic tissue sample obtained by EUS-FNB will be used for FFOCT imaging. The Images will be sent to trained pathologists for diagnosis. The same tissue sample will be sent to the pathology department for routine histological examination. Compare the diagnoses made by the 2 different methods.

SUMMARY:
In most Asian medical centers, rapid on-site cytology evaluation is not available, the number of needle passes of EUS-FNA is decided by endoscopists. Full-field optical coherence tomography (FF-OCT) is a new optical imaging technique that could generate sectioning tomogram from fresh tissue and provide close-to-pathology depiction of the morphological structure and pathological changes in minutes without conventional tissue preparation, slicing, and staining, and dynamic cell imaging (DCI) added the viability information of cells/tissue, which could be more important in sample rapid evaluation.

DETAILED DESCRIPTION:
Light-CT, a special-designed pathology-approximation system which is based on the lighting feature or dynamic feature of tissue and cells, is used to detect malignant cells or tissue in fresh specimens. Morphological structure and pathological changes could be captured in minutes, which implies a possible application in intraoperative diagnosis. The investigators aimed to evaluate the diagnostic efficacy of FFOCT for the tissue samples obtained from EUS-FNB of pancreas.

ELIGIBILITY:
Inclusion Criteria:

* Tissue samples can be obtained via EUS-FNB
* Signed informed consent letter

Exclusion Criteria:

* Unable or refuse to provide informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with pancreatic diseases who receive EUS-FNA/B with tissue sample obtained will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Light-CT | 1week after procedure
  The true positive rate measures the proportion of positives that are correctly identified by Light-CT

SECONDARY OUTCOMES:
Sensitivity of Light-CT | 1week after procedure
  The true negative rate measures the proportion of positives that are correctly identified by Light-CT
The diagnostic efficacy of Light-CT for different pancreatic diseases | 1week after procedure
  Comparing the sensitivity and specificity of FFOCT in the diagnosis of different pancreatic diseases
coherence of FFOCT diagnoses by assistant and pathologist | 1week after procedure
  comparing the diagnostic coherence of FFOCT by trained assistant( endoscopist) and trained pathologist